CLINICAL TRIAL: NCT05662150
Title: Is Low-frequency Repetitive Nerve Stimulation a Reliable Test to Evaluate the Neuromuscular Junction in Myotonic Dystrophy Type 1
Brief Title: Low-frequency Repetitive Nerve Stimulation in Myotonic Dystrophy Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jella De Ville, medical doctor, principal investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Steinert study
Record Dates: First submitted 2022-10-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Questionnaires (Active Comparator): Patients with DM1 were asked to complete a questionnaire to rate a 25-item activity scale (DM1-Activ) and the Myasthenia Gravis Activity of Daily Life scale (MG-ADL) to rate their level of functional burden. For the DM1-Activ a score of 40 alludes no impairment and a score of 0 indicates the highest functional burden of physical activity. This scale has proven to be practical, reliable and valid. For the MG-ADL the total score ranges from 0 to 24, a score of 0 denotes no and 24 the highest functional burden. It should be noted that this scale is not adjusted for DM1. The rationale was to gain information about muscle fatigue and consequently the neuromuscular junction.
  Interventions: Diagnostic Test: Low frequency repetitive stimulation
- grip strength via dynamometer (Active Comparator): The isometric grip strength was tested by using a dynamometer. The subject will be asked to perform an increasing force against the dynamometer over a period of several seconds.
  Interventions: Diagnostic Test: Low frequency repetitive stimulation
- short exercise test (Active Comparator): The subject was asked to contract the ADM muscle as hard as possible in isometric conditions for 10 seconds. CMAP's was recorded 2 seconds after the end of the exercise and then every 10 seconds for 50 seconds.
  Interventions: Diagnostic Test: Low frequency repetitive stimulation
- needle EMG (Active Comparator): The electrical myotonia of each examined muscle was scored according to the Streiss and Sun scale.
  Interventions: Diagnostic Test: Low frequency repetitive stimulation

INTERVENTIONS:
Diagnostic Test: Low frequency repetitive stimulation — Neuromuscular transmission was tested by using short-lasting low frequency RNS (10 stimuli at 3 Hz). The test was applied on the abductor digiti minimi (ADM), anterior tibial, orbiculis oculi, trapezius, anconeus and EDB muscles of one side, in this particular order, by supramaximal stimulation of the corresponding nerve.

SUMMARY:
The study design is a prospective cohort study. It aims to evaluate the neuromuscular junction in dystrophic myotonia 1 (DM 1) using low-frequency repetitive nerve stimulation (RNS) on several nerve-muscle pairs of the one side including proximal and distal muscles of upper and lower extremities. First, it will be investigated whether a decrement with 3 Hz stimulation, as described in literature, is reproducible in our patient population. If this is the case, it will be examined whether it is the consequence of a dysfunction of the neuromuscular junction or rather linked to a hypo-excitability of some muscle fibers due to myotonia. For this purpose, additional tests including short exercise test (to observe any decrement resulting from an inexcitability in myotonic muscle fibers) and needle EMG (for mapping myotonic discharges in the muscles tested with repetitive nerve stimulation) will be performed. Single fiber-EMG will not be provided in this study as an abnormal result does not necessarily indicate a dysfunction of the neuromuscular junction but could just as well be due to the muscular dystrophy in the context of DM1. Finally, it will be investigated if there is a correlation between the decrement

with 3 Hz stimulation and clinical signs as fixed muscle weakness (via Medical Research Counsil (MRC) scale, DM-activ scale [30]) and fatigue (via MG-ADL scale).

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed DM1

Exclusion Criteria:

* minor age
* auto-immune diseases
* medical conditions involving the neuromuscular junction: (myasthenia gravis, Lambert-Eaton myasthenic syndrome, congenital myasthenia syndromes).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Reproducibility of rapid decrement at low frequency stimulation. | 1 year
  Low stimulation frequency was tested in 6 muscles, to verify the presence of an anomalie of the neuromuscular transmission.

SECONDARY OUTCOMES:
Correlation of decrement with grade of EMG-myotonia | 1 year
  Search of correlation between decrement, obtained bij low frequency stimulation, and EMG-myotonia (via needle EMG), to differentiate muscle fiber hypoexcitability in the context of myotonia, from neuromuscular junction block resulting in decrement of the CMA
Is there any clinical expression (muscle fatigability) of a possible neuromuscular junction dysfunction | 1 year
  Search of correlation between muscle fatique (questionnaires and grip strength via dynamometer) and decrement of CMAP (compound muscle action potential).

CONTACTS AND LOCATIONS:
Overall Officials: Jella De Ville, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT05662150/Prot_SAP_000.pdf